CLINICAL TRIAL: NCT00227006
Title: Promoting Long-term Dietary Change to Reduce CVD Risk
Brief Title: Promoting Long-term Behavior Change to Reduce CVD Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Unrestricted research gift from Nutrilite Health Institute (Unknown)
Responsible Party: Principal Investigator, Michaela Kiernan, Senior Research Scientist, Stanford University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: R29HL060154 (NIH); R29HL060154 (NIH); NCT00005747 (obsolete NCT alias)
Record Dates: First submitted 2005-09-13; First posted 2005-09-27 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- Taste-Based Goal Setting (Experimental): 6-month intervention (14 lifestyle counseling classes)
  Interventions: Behavioral: Behavioral lifestyle/weight-loss intervention
- Smart Consumers (Active Comparator): 6-month intervention (14 lifestyle counseling classes)
  Interventions: Behavioral: Behavioral lifestyle/weight-loss intervention
- Community Access (Active Comparator): Can enroll in behavioral treatment programs available in the community that do not include medication or very-low calorie diets
  Interventions: Behavioral: Behavioral lifestyle/weight-loss intervention

INTERVENTIONS:
Behavioral: Behavioral lifestyle/weight-loss intervention

SUMMARY:
Once intervention class or staff contact is removed, obese adults participating in behavioral weight-loss programs often give up healthy eating habits and regain weight. We examined whether taste-based goal setting, which minimizes perceived deprivation by promoting taste and moderation, would sustain long-term reductions in saturated fat and body mass index (BMI).

DETAILED DESCRIPTION:
Once intervention class or staff contact is removed, obese adults participating in behavioral weight-loss programs often give up healthy eating habits and regain weight. We examined whether taste-based goal setting, which minimizes perceived deprivation by promoting taste and moderation, would sustain long-term reductions in saturated fat and body mass index (BMI). Participants were randomized to Taste-Based Choices (taste-based goal setting + a standard 6-month behavioral weight-loss intervention), Smart Consumers (a standard 6-month intervention alone) or Community Access (access to commercial/community-based behavioral weight-loss programs) and followed over 18 months. To test our hypotheses, we examined a set of orthogonal contrasts (TBC and SC vs. CA; TBC vs. SC) on reductions in saturated fat (Block FFQ) and clinic-measured BMI.

ELIGIBILITY:
Inclusion Criteria:- Body mass index between 27-37

* Physically inactive
* Able to participate in physical activity
* Percentage of daily calories from total fat 30% or more
* Free of diagnosed heart disease
* Stable on medications for 3 months or more Exclusion Criteria:- Diabetic
* Dysphoric (Beck Depression Inventory score greater than 18)
* Binge eating or bulimic (Eating Disorder Diagnostic Scale)

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 1999-01; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Percentage of saturated fat in diet | 18 months

SECONDARY OUTCOMES:
Body weight | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Michaela Kiernan, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Background] Goldberg JH, Kiernan M. Innovative techniques to address retention in a behavioral weight-loss trial. Health Educ Res. 2005 Aug;20(4):439-47. doi: 10.1093/her/cyg139. Epub 2004 Dec 14. PMID 15598664
- [Background] Kraemer HC, Kiernan M, Essex M, Kupfer DJ. How and why criteria defining moderators and mediators differ between the Baron & Kenny and MacArthur approaches. Health Psychol. 2008 Mar;27(2S):S101-8. doi: 10.1037/0278-6133.27.2(Suppl.).S101. PMID 18377151